CLINICAL TRIAL: NCT05946421
Title: The BASA Study: Breath Analysis for Severe Asthma Patients. A New, Non-invasive Approach for the Monitoring of Inflammation in Severe Asthma Patients on Biologics
Brief Title: The BASA Study: Breath Analysis for Severe Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Stefania Principe, MD, PhD, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Other Study IDs: Università di Palermo
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Severe Asthma
Keywords: severe asthma; exhaled breath; biologics; monitoring
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Asthma patients on biologics
  Interventions: Device: exhaled breath analysis
- Healthy controls
  Interventions: Device: exhaled breath analysis

INTERVENTIONS:
Device: exhaled breath analysis — non invasive technology to measure components of exhaled breath

SUMMARY:
This study will evaluate the fluctuations of exhaled breath markers in patients with severe asthma on biologics. In the study, severe asthma patients will be followed up to 16 weeks monitoring lung function and inflammation through non-invasive technologies such as exhaled breath analysis (FeNO, GC-MS and EBC). A control group will be followed up to two weeks with the overall objective to indentify and evaluate the modifcations of markers of inflammation in patient under biologic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma diagnosis according to the latest recommendation
* Eligible or in treatment with a biologic treatment for severe asthma
* Able to follow istructions
* Able and willing to sign the informed consent

Exclusion Criteria:

* Not able to perform lung function measurements and the procedures of the study
* Acute respiratory or non respiratory infection (<4 weeks)
* Not willing to continue the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe asthma patients eligible or already on biologic treatment that are able to follow regular visits at 2, 4, 8, 16 weeks, and to perform lung function and exhaled breath analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-02-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the fluctuations of markers of inflammation in patients with severe asthma under biologic therapy | 16 weeks

SECONDARY OUTCOMES:
evaluate whether the measurement of H2O2 could be considered as a marker of inflammation in severe asthma patients | 16 weeks

OTHER OUTCOMES:
evaluate whether there are specific exhaled biomarkers useful to monitor patients with severe asthma on long-term treatment with biologics | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AOUP Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Undecided